CLINICAL TRIAL: NCT00518739
Title: A Phase I Dose Escalation Study of MK2461 in Patients With Advanced Cancer
Brief Title: MK2461 in Patients With Advanced Cancer (2461-001)(COMPLETED)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2461-001; 2006_530
Record Dates: First submitted 2007-08-17; First posted 2007-08-21 (Estimated); Last update posted 2015-03-27 (Estimated); Status verified 2015-03

CONDITIONS: Advanced Cancer
MeSH Terms: interventions — 5H-benzo(4,5)cyclohepta(1,2-b)pyridin-5-one

INTERVENTIONS:
Drug: MK2461 — Patients will be administered oral MK2461 twice daily and will be treated for 28 day cycles. Patients will be enrolled in cohorts and will be treated at sequentially rising dose levels of MK2461. 60 mg dry filled capsules, escalating to 240 mg ( for dosing in Cohort 4 & beyond).

SUMMARY:
This is a first-in-human trial to establish the safety, tolerability, Recommended Phase II Dose (RP2D), pharmacodynamic, and clinical activity of MK2461.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age, with adequate organ function, and an ECOG performance of <2
* Patients must be willing to undergo pre-study and post dose tumor biopsy and have tumor accessible to biopsy (waived during Part A)

Exclusion Criteria:

* No chemotherapy, radiotherapy, or biological therapy with 4 weeks of study participation
* Patients must not have primary central nervous system tumor
* Patient has had prescription or non-prescription drugs or other products known to be metabolized by CYP3A4 that cannot be discontinued prior to Day 1 of dosing and withheld throughout the study until 2 weeks after the last dose of study medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2007-02; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and tolerability of MK2461 | 18 Months

SECONDARY OUTCOMES:
To determine the Recommend Phase II Dose or doses (RP2D) based on safety, tumor pharmacodynamics, and parmacokinetics. | 18 Months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC